CLINICAL TRIAL: NCT01303224
Title: Double-blind, Randomised, Placebo-controlled, Parallel-group Phase II Study to Evaluate the Effect of Oral Ibodutant in Irritable Bowel Syndrome With Diarrhoea (IBS-D).
Brief Title: Ibodutant for Relief of Irritable Bowel Syndrome With Diarrhoea (IBS-D)
Acronym: IRIS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAK-04; 2010-018300-85 (EudraCT Number)
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Results first posted 2013-03-25 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-09

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; Colon, irritable; Bowel disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Intestinal Diseases | interventions — ibodutant; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibodutant low dose (Experimental): Oral tablet, to be given once daily in fasting conditions.
  Interventions: Drug: Ibodutant
- Ibodutant intermediate dose (Experimental): Oral tablet, to be given once daily in fasting conditions.
  Interventions: Drug: Ibodutant
- Ibodutant high dose (Experimental): Oral tablet, to be given once daily in fasting conditions.
  Interventions: Drug: Ibodutant
- Placebo (Placebo Comparator): Oral tablet, to be given once daily in fasting conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibodutant — Oral tablet, low dose, once daily, for 8 weeks
  Other Names: Code: MEN 15596
  Arms: Ibodutant low dose
Drug: Ibodutant — Oral tablet, intermediate dose, once daily, for 8 weeks
  Other Names: Code: MEN 15596
  Arms: Ibodutant intermediate dose
Drug: Ibodutant — Oral tablet, high dose, once daily, for 8 weeks
  Other Names: Code: MEN 15569
  Arms: Ibodutant high dose
Drug: Placebo — Oral tablet, (identical in appearance and weight to Ibodutant tablets), once daily, for 8 weeks
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome with diarrhoea (IBS-D) is a functional gastrointestinal disorder characterised by chronic or recurrent abdominal pain or discomfort and diarrhoea. This trial aims at the evaluation of the efficacy and safety of the neurokinin type 2 receptor antagonist Ibodutant in improving IBS-D symptoms.

DETAILED DESCRIPTION:
The study evaluates the efficacy and safety of three doses of ibodutant, given once daily for 8 weeks versus placebo in IBS-D patients. Efficacy is evaluated in terms of overall symptom relief and abdominal pain/discomfort relief after 8 weeks of treatment. The clinical phase of the study comprises a 2-week run-in period (treatment-free),an 8-week double-blind treatment period and a 2-week treatment withdrawal period, resulting in a 10-week overall duration of the study for each patient.

Patients report their IBS-related symptoms daily in an electronic diary (web-and telephone based)during all periods of the study.

ELIGIBILITY:
Inclusion Criteria:

At start of the run-in period:

* Male or female patients aged 18 - 70 years with a clinical diagnosis of IBS-D according to the Rome III criteria:
* Recurrent abdominal pain/discomfort for at least 3 days per month in the last 3 months associated with at least 2 of the following characteristics:

  1. improvement with defecation;
  2. onset associated with a change in the frequency of stool;
  3. onset associated with a change in form (appearance) of stool.
* Symptom-onset at least 6 months prior to diagnosis.
* Loose/watery stools at least 25% of the time in the last 3 months AND hard/lumpy stools less than 25% of the time in the last 3 months.
* More than 3 bowel movements per day at least 25% of the time in the last 3 months.
* For patients older than 50 years OR patients with positive family history of colorectal cancer: Normal results from colonoscopy or flexible sigmoidoscopy.
* Mentally competent, able to give written informed consent.
* For women of childbearing potential: Use of a highly effective contraceptive method throughout the entire study period and up to 30 days post-treatment.
* Normal physical examination or without clinically relevant abnormalities.

At randomisation:

-Confirmation of IBS-D severity in terms of bowel movement frequency and abdominal pain intensity along the 2-week run-in period.

Exclusion criteria:

* Organic abnormalities of the gastrointestinal tract, including history of colonic or major abdominal surgery.
* History of gluten enteropathy.
* Lactose intolerance as assessed by response to diet.
* History of positive tests for ova or parasites, or occult blood in the stool.
* Previous diagnosis of diabetes mellitus (either type 1 or 2).
* Unstable medical condition.
* Major psychiatric, neurological, or cardiovascular disorders, or uncontrolled metabolic disease.
* Relevant changes in dietary habits, lifestyle, or exercise regimen in the previous 2 months.
* Use of concurrent medication with drugs known to interfere with gastro-intestinal motility or sensitivity.
* Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Study Chair — Department of Gastroenterology, University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium
Locations (71):
- Bulgaria (10):
  - MHAT "Haskovo", Second Internal Department, Haskovo
  - UMHAT "Dr. Georgi Stranski", Clinic of Gastroenterology, Pleven
  - MHAT "Kaspela", Department of Gastroenterology, Plovdiv
  - UMHAT "Sveti Georgi", Internal Consultative Department, Plovdiv
  - MHAT "Ruse", Clinic of Gastroenterology, Rousse
  - Fifth City Hospital, Gastroenterology Department, Sofia
  - UMHAT "Alexandrovska", Clinic of Propedeutic of Internal Disease, Sofia
  - MHAT "Sveta Anna", Department of Gastroenterology, Endocrinology, and Nephrology, Sofia
  - UMHAT "St. Marina", Clinic of Gastroenterology, Varna
  - MHAT "Dr. Stefan Cherkezov", Gastroenterology Department, Veliko Tarnovo
- Czechia (7):
  - Poliklinika III, Hepato-Gastroenterologie HK, Hradec Králové
  - Gastromedic s.r.o., Soukroma ordinace, Pardubice
  - IKEM, Klinika hepatogastroenterologie, Prague
  - Hospital Slany, Internal Department, Slaný
  - District Hospital, Internal Department, Strakonice
  - Regional Hospital Tabor, Gastroenterology, Tábor
  - Kojecký Soukroma Ordinace, Zlín
- Denmark (5):
  - CCBR Aalborg, Aalborg
  - CCBR Ballerup, Ballerup Municipality
  - Gentofte Hospital, Medicinsk Afdeling F, Hellerup
  - Regionshospitalet Silkeborg, Medicinsk Afdeling F, Silkeborg
  - CCBR Vejle, Vejle
- Germany (8):
  - Klinische Forschung Berlin, Berlin
  - Universitätsklinik Köln, Gastroenterologie, Cologne
  - ABX-CRO Clinical Research GmbH, Dresden
  - Private Practice Dr. Schaefer, Essen
  - Clinical Research Hamburg, Hamburg
  - Israelitisches Krankenhaus, Innere Medizin, Hamburg
  - Gemeinschaftspraxis Kuchta, Wegner, Schiefke, Leipzig
  - Praxis Prof. Kellner, Munich
- Italy (9):
  - Ospedale Valduce, Unità Operativa Complessa di Gastroenterologia, Como
  - Azienda Ospedaliera Sant'Anna, U.O. Di Gastroenterologia, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, USOD Gastroenterologia 1, Florence
  - Università degli Studi di Genova, Dipartimento di Medicina Interna e Specialità Mediche, Genoa
  - Azienda Ospedaliera - Università di Padova, Struttura Operativa Complessa di Gastroenterologia, Padua
  - IRCCS Policlinico San Matteo, Dipartimento di Medicina Interna I e Gastroenterologia, Pavia
  - "Ospedale Nuovo Santa Chiara-Cisanello, Dipartimento di Medicina Interna, Pisa
  - IRCCS Istituto Clinico Humanitas, Dipartimento di Gastroenterologia, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, Divisione di Gastroenterologia, San Giovanni Rotondo
- Poland (18):
  - NZOZ Specjalistyczne Centrum Gastrologii "Gastromed", Bialystok
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Gabinet Lekarski Janusz Rudziński, Bydgoszcz
  - Mazowieckie Centrum Badań Klinicznych I.Czajkowska M.Śmietańska s.c., Grodzisk Mazowiecki
  - Specjalistyczne Centrum Medyczne "NOWOMED", Krakow
  - 5 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ w Krakowie, Krakow
  - NZOZ Krakowskie Centrum Medyczne, Krakow
  - Instytut Medycyny Wsi im. Witolda Chodźki Publiczny Zakład Opieki Zdrowotnej, Lublin
  - NZOZ "Centrum Alergologii", Lublin
  - NZOZ Solumed, Poznan
  - NZOZ Zaspół Poradni Specjalistycznych "Artmed", Poznan
  - Endoskopia Sp. z o.o., Sopot
  - NZOZ "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych, Torun
  - NZOZ Remedis Sp z o.o., Torun
  - Centrum Badawcze Współczesnej Terapii, Prywatny Gabinet Lekarski, Warsaw
  - Centrum Medyczne "Osteomed" Sp. z o. o, Warsaw
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - NZOZ Vivamed, Warsaw
- Spain (8):
  - Hospital Germans Trias i Pujol, Digestive Unit, Badalona
  - Centro Medico Teknon, Gastroenteloroly Service, Barcelona
  - "Hospital Universitario Virgen de la Arrixaca, Servicio de Medicina del Aparato Digestivo, El Palmar (Murcia)
  - Hospital Clinico San Carlos, Digestive Diseases, Madrid
  - Hospital de Mataró, Unitat d'Exploracions Funcionals Digestives, Mataró
  - Corporació Sanitària Parc Tauli, Sabadell
  - Complejo Hospitalario Universitario de Santiago, Gastroenterology, Santiago de Compostela
  - Hospital Virgen Macarena, Digestive Service, Seville
- Sweden (6):
  - Sahlgrenska Universitetssjukhuset, Mag-tarm lab, Gothenburg
  - Probare, Lund
  - Clinical Research Support, S-huset, Södra Grev Rosengatan, Örebro
  - Kärnsjukhuset, Skövde
  - Gastrocentrum Aleris specialistvård Sabbatsberg,, Stockholm
  - Akademiska sjukhuset, Gastromottagningen, Uppsala

REFERENCES:
- [Derived] Tack J, Schumacher K, Tonini G, Scartoni S, Capriati A, Maggi CA; Iris-2 investigators. The neurokinin-2 receptor antagonist ibodutant improves overall symptoms, abdominal pain and stool pattern in female patients in a phase II study of diarrhoea-predominant IBS. Gut. 2017 Aug;66(8):1403-1413. doi: 10.1136/gutjnl-2015-310683. Epub 2016 Apr 15. PMID 27196574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject screened 06/10/2010, first subject randomised 22/10/2010, last subject out 11/05/2012, at 78 study sites in 8 European countries (Bulgaria, Czech Republic, Denmark, Germany, Italy, Poland, Spain, and Sweden)
Pre-assignment Details: A run-in period was planned to confirm eligibility criteria. 5 more patients were randomized instead of the planned number (560) because due to the high screen fail rate it was impossible to predict with how many patients the enrollment goal would be reached. Although the enrollment goal was reached these 5 patients in screening continued the study
Groups:
- Ibodutant 1 mg; Ibodutant 3 mg; Ibodutant 10 mg; Placebo: oral tablet, once daily
Period: Overall Study
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Started | 141 (randomised, safety population, >= 1 dose of study medication) | 142 (randomised, safety population, >= 1 dose of study medication) | 139 (randomised, safety population, >= 1 dose of study medication) | 143 (randomised, safety population, >= 1 dose of study medication)
Intention To Treat | 140 (subjects with at least 1 primary endpoint evaluation post randomisation) | 138 (subjects with at least 1 primary endpoint evaluation post randomisation) | 139 (subjects with at least 1 primary endpoint evaluation post randomisation) | 142 (subjects with at least 1 primary endpoint evaluation post randomisation)
Completed | 130 | 131 | 133 | 133
Not Completed | 11 | 11 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo | Total
Number analyzed (Participants) | 140 | 138 | 139 | 142 | 559
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.7) | 47.1 (13.4) | 47.0 (12.8) | 44.1 (14.0) | 46.0 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 87 | 79 | 78 | 333
  Male | 51 | 51 | 60 | 64 | 226
Time since onset of IBS symptoms [Mean (Standard Deviation); unit: years] | 6.2 (7.3) | 6.3 (7.5) | 6.3 (6.9) | 4.6 (6.2) | 5.8 (7.0)
IBS symptoms at baseline/ randomisation) [Mean (Standard Deviation); unit: Scores on a scale] — 5 point scale ranging from "0"= no symptoms to "4"= very severe
  Scores on a scale
    Abdominal pain score | 2.5 (0.6) | 2.3 (0.5) | 2.3 (0.5) | 2.3 (0.6) | 2.3 (0.5)
    Bloating score | 2.4 (0.8) | 2.2 (0.7) | 2.2 (0.7) | 2.2 (0.6) | 2.3 (0.7)
    Urgency score | 2.5 (0.7) | 2.5 (0.6) | 2.4 (0.6) | 2.4 (0.6) | 2.4 (0.7)
    IBS symptom severity rate | 2.7 (0.7) | 2.6 (0.6) | 2.6 (0.6) | 2.6 (0.6) | 2.7 (0.6)
Stool frequency/day [Mean (Standard Deviation); unit: bowel movements/day] — Overall stool frequency per day
  bowel movements/day | 4.6 (1.5) | 4.4 (1.3) | 4.4 (1.5) | 4.4 (1.2) | 4.5 (1.4)
Stool consistency [Mean (Standard Deviation); unit: Scores on a scale] — 7-point Bristol stool scale ranging from "1"= hard lumpy stool to "7"= watery, liquid stool
  Scores on a scale | 5.7 (0.6) | 5.7 (0.5) | 5.7 (0.6) | 5.7 (0.6) | 5.7 (0.6)
IBS-Symptom Severity Scale score [Mean (Standard Deviation); unit: Scores on a scale] — IBS symptom severity score, ranging from "0"= no symptoms to "500"= very severe symptoms
  Scores on a scale | 343.4 (68.8) | 333.3 (78.3) | 332.6 (74.3) | 335.7 (69.4) | 336.3 (72.7)
European Quality of Life Questionnaire 5D (EQ-5D) QoL VAS [Mean (Standard Deviation); unit: Scores on a scale] — European quality of life visual analogue scale ranging from "0"= worst imaginable health state to "100"= best imaginable health state
  Scores on a scale | 54.5 (22.9) | 55.5 (21.9) | 58.1 (22.9) | 55.3 (22.3) | 55.8 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Response for Relief of Overall IBS Symptoms and of Abdominal Pain/Discomfort at the End of 8 Weeks of Treatment, Where the Response is Defined as at Least 6 Weeks With Satisfactory Relief During 8 Weeks of Treatment (75% Rule); Intention-to-treat (ITT).
Description: Weekly binary questions (yes/no) from Interactive Voice/Web Response (IV/WRS) diary records: "Did you have satisfactory relief of your overall IBS symptoms during the last week?" and "Did you have satisfactory relief of your abdominal pain or discomfort during the last week?"
  Responder: Report of satisfactory overall IBS symptom relief ="Yes" and of satisfactory abdominal pain/discomfort relief = "Yes" 6/8 weeks (75% rule)
Time Frame: Eight weeks
Population: Intention-to-Treat (559)
Measure: Number; unit: participants
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 140 | 138 | 139 | 142
participants
  Responders according to the 75% rule/"Yes" | 45 | 46 | 55 | 39
  Responders according to the 75% rule/"No" | 95 | 92 | 84 | 103
Statistical Analysis 1: Comparison: Ibodutant 1 mg vs Ibodutant 3 mg vs Ibodutant 10 mg vs Placebo; Mantel-Haenszel-Test was used to compare separately each of the 3 active treatment groups with placebo using a two-sided overall significance level of 5%. The proportion of responders was tested with the following hypotheses: H0 (placebo) vs H1(Ibodutant:1mg/3mg/10mg). Approximately 80% power based on the assumptions: rate placebo 40%, expected mean therapeutic gain over placebo 15% for at least one dose of Ibodutant; Test type: Superiority or Other; p < 0.05, Mantel Haenszel — Multiplicity was adjusted by using the Hochberg Procedure

2. Secondary Outcome: Response for Relief of Overall IBS Symptoms and of Abdominal Pain/Discomfort at the End of 8 Weeks of Treatment, Where the Response is Defined as at Least 4 Weeks With Satisfactory Relief During 8 Weeks of Treatment (50% Rule) in the ITT Population
Description: Weekly binary questions (yes/no) from IV/WRS diary records: "Did you have satisfactory relief of your overall IBS symptoms during the last week?" and "Did you have satisfactory relief of your abdominal pain or discomfort during the last week?"
  Responder: Report of satisfactory overall IBS symptom relief ="Yes" and of satisfactory abdominal pain/discomfort relief = "Yes" 4/8 weeks with at least 2 consecutive weeks of satisfactory relief during Week 5 to Week 8(50% rule)
Time Frame: Eight weeks
Population: Intention-to-Treat (559)
Measure: Number; unit: participants
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 140 | 138 | 139 | 142
participants
  Responders according to the 50% rule/"Yes" | 72 | 61 | 74 | 55
  Responders according to the 50% rule/"No" | 68 | 77 | 65 | 87
Statistical Analysis 1: Comparison: Ibodutant 1 mg vs Ibodutant 3 mg vs Ibodutant 10 mg vs Placebo; Test type: Superiority or Other; p < 0.05, Mantel Haenszel — Multiplicity was adjusted using the Hochberg procedure

3. Secondary Outcome: Quality of Life Changes (Using EuroQoL EQ-5D Questionnaire)
Description: Change in EQ-5D Quality of Life (visual analogue scale) score at the end of 8 weeks of treatment versus baseline (at randomisation). EQ-5D quality of life visual analogue scale ranges from "0"= worst imaginable health state to "100"=best imaginable health state.
Time Frame: Eight weeks
Population: Intention-to-treat; i.e. all ITT patients who provided EQ-5D data at Visit 2 (start of treatment) and Visit 4 (end of treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 131 | 133 | 133 | 131
units on a scale
  Baseline (randomisation) | 56.4 (20.6) | 58.2 (22.0) | 57.2 (22.0) | 58.7 (21.5)
  Visit 4 | 71.3 (17.2) | 72.1 (18.7) | 66.7 (20.7) | 72.2 (17.0)

4. Other Pre Specified Outcome: Subgroup Analysis: Response for Relief of Overall IBS Symptoms and of Abdominal Pain/Discomfort According to the 75% Rule in the Female ITT Population
Description: Weekly binary questions (yes/no) from IV/WRS diary records: "Did you have satisfactory relief of your overall IBS symptoms during the last week?" and "Did you have satisfactory relief of your abdominal pain or discomfort during the last week?"
  Responder: Report of satisfactory overall IBS symptom relief ="Yes" and of satisfactory abdominal pain/discomfort relief = "Yes" 6/8 weeks (75% rule)
Time Frame: Eight weeks
Population: Intention-to-Treat in the female population (333)
Measure: Number; unit: participants
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 89 | 87 | 79 | 78
participants
  Responders according to 75% rule/"Yes" | 32 | 35 | 37 | 19
  Responders according to 75% rule/"No" | 57 | 52 | 42 | 59

5. Other Pre Specified Outcome: Subgroup Analysis: Response for Relief of Overall IBS Symptoms and of Abdominal Pain/Discomfort According to the 75% Rule in the Male ITT Population
Description: as for outcome 4
Time Frame: Eight weeks
Population: Intention-to-Treat in the male population (226)
Measure: Number; unit: participants
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Number analyzed (Participants) | 51 | 51 | 60 | 64
participants
  Responders according to the 75% rule/"Yes" | 13 | 11 | 18 | 20
  Responders according to the 75% rule/"No" | 38 | 40 | 42 | 44

ADVERSE EVENTS:
Time Frame: 8 weeks for Treatment Emergent Signs and Symptoms (TESS)
Description: TESS (collected from first drug intake at Visit 2 (randomisation) during the treatment period of 8 weeks) were analysed for the Safety Population (all patients who took at least one dose of study medication, N = 565).
  Generally, Adverse Events were reported/patient for a period of 12 weeks (during the total individual study period).
Arm/Group | Ibodutant 1 mg | Ibodutant 3 mg | Ibodutant 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/141 | 1/142 | 1/139 | 3/143
Other Adverse Events (participants affected / at risk) | 20/141 | 19/142 | 29/139 | 20/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 1 mg (N=141) | Ibodutant 3 mg (N=142) | Ibodutant 10 mg (N=139) | Placebo (N=143)
Mydriasis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes Mellitus type II (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsened Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterus Myomatosus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 1 mg (N=141) | Ibodutant 3 mg (N=142) | Ibodutant 10 mg (N=139) | Placebo (N=143)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (6) | 4 (4) | 5 (5) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 3 (3) | 8 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the PI will allow Sponsor at least 60 days time to review and comment upon the publication manuscript. No publication of PI is permitted before the overall publication of the multicentre study made by the Sponsor (or its designee), unless said overall publication is not made within 18 months from the completion of the Final Study Report.